CLINICAL TRIAL: NCT05899062
Title: Investigation of the Effect of Telerehabilitation-based Exercise Training on Constipation Symptoms and Quality of Life.
Brief Title: Telerehabilitation-based Exercise Training in Constipated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Raziye Şavkın, Assoc. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-60116787-020-309406
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2023-06

CONDITIONS: Constipation
Keywords: Constipation; Telerehabilitation; Exercise; Quality of life; Constipation symptoms
MeSH Terms: conditions — Constipation; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): The patients in the control group will be given education about constipation, which lasts about 45-60 minutes, with the telerehabilitation method. In addition, a "Constipation Training Booklet" will be sent via e-mail or WhatsApp, related to the training content given to all patients and to reinforce the training. Definition of constipation in education, its causes, medications that cause constipation, risk factors, suggestions for prevention of constipation (such as regular defecation, not delaying defecation, best position for defecation, not straining for a long time), constipation treatment and the importance of individual management, healthy and balanced diet, nutrition Types, adequate fluid intake, benefits of exercise and appropriate exercise selection, abdominal massage, toilet training and individual methods of preventing constipation will be included.
  Interventions: Other: Education with the telerehabilitation method. In addition, a "Constipation Training Booklet" will be sent via e-mail or WhatsApp
- Intervention group (Other): The patients in intervention group will be given an exercise program in addition to all the practices in the control group. Training and exercise practices will be carried out with the telerehabilitation method. Exercise training, which will last 40-60 minutes, 3 days a week for 4 weeks, will consist of warm-up and breathing exercises, exercises for constipation and cooling movements. Patients will be asked to walk for at least 30 minutes, 2 days a week, on days without exercise training.
  Interventions: Other: Training and exercise practices with the telerehabilitation method.

INTERVENTIONS:
Other: Education with the telerehabilitation method. In addition, a "Constipation Training Booklet" will be sent via e-mail or WhatsApp — The patients in the control group will be given education about constipation, which lasts about 45-60 minutes, with the telerehabilitation method. In addition, a "Constipation Training Booklet" will be sent via e-mail or WhatsApp, related to the training content given to all patients and to reinforce the training. Definition of constipation in education, its causes, medications that cause constipation, risk factors, suggestions for prevention of constipation (such as regular defecation, not delaying defecation, best position for defecation, not straining for a long time), constipation treatment and the importance of individual management, healthy and balanced diet, nutrition Types, adequate fluid intake, benefits of exercise and appropriate exercise selection, abdominal massage, toilet training and individual methods of preventing constipation will be included.
  Arms: Control group
Other: Training and exercise practices with the telerehabilitation method. — The patients in this group will be given an exercise program in addition to all the practices in the control group. Training and exercise practices will be carried out with the telerehabilitation method. Exercise training, which will last 40-60 minutes, 3 days a week for 4 weeks, will consist of warm-up and breathing exercises, exercises for constipation and cooling movements. Patients will be asked to walk for at least 30 minutes, 2 days a week, on days without exercise training.
  Arms: Intervention group

SUMMARY:
It has been determined that three out of every four people in the society do not have sufficient physical activity level, and 54% of individuals between the ages of 15-19 and over 55 are sedentary. As a result of this, the probability of encountering the problem of constipation may increase. There are many methods in the treatment of constipation. When examined in terms of exercise interventions, it was found that 150 minutes of moderate-intensity exercise per week was effective in reducing the symptoms of constipation, while aerobic exercise performed less than 140 minutes/week did not improve the symptoms of constipation. It has been reported that individuals who received defecation training were particularly successful in the management of constipation symptoms.

In our study, it is aimed to examine the effectiveness of exercise interventions for constipation. In addition, to the best of our knowledge, no study has been conducted on the effectiveness of a telerehabilitation-based education and exercise program in patients with constipation. It is thought that the management of patients with constipation with telerehabilitation will ease the burden on the health system, while it will save the patient cost and time, and will facilitate the access to treatment for patients living in geographically disadvantaged areas. In addition, it is important for patients to participate in distance rehabilitation studies in their professional and social lives, as it is an innovative treatment approach. It is thought that the exercises for constipation applied in addition to the training program may be a more effective method in improving the quality of life and colonic motility of the patients.

DETAILED DESCRIPTION:
Constipation is the problem of insufficient defecation caused by individual factors and is defined as less than three defecations per week according to health professionals. In chronic constipation, decreased frequency of defecation, hard stool, feeling of incomplete excretion of feces and straining are seen. From a biopsychosocial point of view, it negatively affects the health-related quality of life of the individual and is a health problem seen at a high rate in the society (Lembo and Camilleri 2003, Talley 2004). This situation is seen as a result of aging and affects women 2-3 times more than men (Huang et al. 2017). The incidence of constipation is seen at a rate of 22-40% in our country, in other nations is seen at a rate varies between 2 and 34%. (Kasap and Bor 2006, Uysal et al. 2010). Its etiology is multifactorial; It may occur as a result of metabolic disorders, drugs used, stress, perianal dysfunctions and other reasons (Heidelbaugh et al. 2021).

While pharmacological treatment agents such as laxatives, chlorine channel activators and osmotic agents are used in the treatment of chronic constipation, lifestyle recommendations including diet, probiotics and physical activity are also used. In some chronic cases, surgical methods are preferred (Leung et al. 2011). Some of the physiotherapy interventions used in the management of constipation are: Biofeedback, tens, interference flow and exercise (LaCross et al. 2022). It is reported that especially exercise is effective in reducing the symptoms of constipation (Gao et al. 2019).

In a study examining the effects of exercise and patient education on constipation, it was reported that regular walking for 20-30 minutes a day for 12 weeks could improve constipation symptoms (Yi et al. 2014). It has been found that 150 minutes of moderate-intensity exercise per week is effective in reducing constipation symptoms, while aerobic exercise performed less than 140 minutes/week does not reduce symptoms of constipation (De Schryver et al. 2005). It is also reported that individuals who receive defecation training are successful in managing their constipation symptoms (Ruitong Gao et al. 2019). Therefore, it is thought that lifestyle education and exercise may be effective in the management of constipation symptoms.

It has been specified that three out of every four people in the society do not have sufficient physical activity level, and especially 54% of individuals between the ages of 15-19 and over 55 are sedentary. This sedentary lifestyle and decreased physical activity may cause constipation by negatively affecting the colonic transit time (Active Living Association 2010, De Schryver et al. 2005). It has been reported that the exercise and nutrition program reduces the use of laxatives while eliminating the symptoms of constipation in patients (Ceren Orhan et al 2015). Similarly, daily moderate-intensity exercise was found to reduce constipation symptoms by 44% in women (Dukas et al. 2033).

Lack of exercise may predispose the individual to neurological diseases or musculoskeletal disorders. As a result, symptoms of abdominopelvic dyssynergia and constipation occur over time. In the treatment, it is aimed to optimize the motor coordination of the abdominal and anal muscles (Wilson 2020, Grimes 2022). Physiotherapists are effective in organizing the muscles and directing the internal pressure with the help of exercise methods in these dysfunctions. Thus, colonic transition is facilitated; while the rectum contracts, the anal sphincters can relax in time (De Schryver et al 2005).

In addition, the use of exercise programs that provide vibration in the abdominal region can cause contractions in the abdominal muscles.It is thought that this may be effective in reducing the symptoms of constipation by inducing colonic movements (Peters HP and De Vries 2001).

Physiotherapy and rehabilitation interventions, especially exercise therapy, are recommended in the treatment of constipation. However, individuals who live in remote or rural areas or cannot allocate time for such treatments due to factors such as working conditions, workplace permission problems, time and distance may find it difficult to access treatment. A possible solution in this context is to provide remote rehabilitation services with the help of telerehabilitation technology (Russell 2009). Telerehabilitation is the provision of remote rehabilitation service with the help of digital technology. Through such services, education can be provided to the patients and family members. In addition, telerehabilitation may include patient evaluation, diagnosis, treatment and follow-up of the prognosis. Thanks to tele-rehabilitation, patients living in geographically disadvantaged areas have the opportunity to access rehabilitation. As a result, the burden on the health system is reduced and time and transportation costs are saved for the patient.It may also provide additional benefits related to rehabilitation in patients' own occupational and social environments (Russell et al. 2011). As far as investigators know, there is no study on telerehabilitation enforcement in the management of constipation in the literature.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old,
* Diagnosed with constipation
* Fewer than three defecations per week
* Straining in more than 25% of defecations
* Lumpy or hard stools in more than 25% of defecations
* Sensation of incomplete emptying of stool in more than 25% of defecations
* More than 25% of defecations have a feeling of being stuck or blocked
* Requirement of manual maneuvering to facilitate at least 25% of defecations (e.g. finger emptying, support of the pelvic floor muscles)
* Rarely loose stools without the use of laxatives
* Those who have insufficient criteria for irritable bowel syndrome,
* Being sedentary (doing 30 minutes or less of moderate physical activity most days of the week),
* Those who have not participated in diet control/weight reduction programs in the last 6 months,
* To be able to understand, speak and write Turkish,
* To be able to understand the verbal and written information given,
* Having internet access,
* To be able to use video conferencing software.

Exclusion Criteria:

* Those who use drugs that affect defecation other than laxatives,
* Patients who have had previous digestive system surgery,
* Those who will undergo abdominal surgery,
* Those who have undergone major surgery in the abdominal and perianal region,
* Those with congenital megacolon, pseudoobstruction and anorectal disease,
* Those with any orthopedic limitations,
* Those with comorbid diseases such as cancer,
* Those with neurological diseases that cause functional disability,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Form Scale | 2 Minutes
  Visual sampling is used to obtain information about the consistency, thickness and amount of stool by specifying 7 different types of stool. In this way, rough information about both bowel work and defecation function is obtained.

SECONDARY OUTCOMES:
Constipation Assessment Scale | 5 Minutes
  This scale is a constipation assessment scale consisting of 8 items. Each item is given a score between 0-2. The total score of the scale is obtained by summing the scores from all items. A score of 0 indicates the absence of constipation, and a score of 16 indicates the presence of severe constipation. The higher the score, the higher the severity of constipation.

OTHER OUTCOMES:
Constipation Severity Scale (CSS) | 10 Minutes
  This scale is used in determining the problem of constipation and grading its severity. There are 16 questions in total within the scope of the scale. CCS includes Large Intestine Laziness, Stool Obstruction and Pain sub-dimension. Scores range from 0 to 29 in the Large Intestine Laziness dimension, between 0 and 28 in the Fecal Obstruction dimension, and between 0 and 16 in the Pain dimension. In this context, the lowest score that can be obtained is 0, while the highest score is 73. The high scores obtained from the scale indicate that the symptoms are at a serious level.
Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire | 10 Minutes
  It was developed to assess the effects of chronic constipation on quality of life and activities of daily living, and the severity of constipation symptoms. Items are scored on 5-point Likert scales ranging from 0 to 4 (0 = 'no symptoms', 1 = 'mild', 2 = 'moderate', 3 = 'severe', and 4 = 'very severe'). An average total score in the range of 0-4 is obtained by dividing the total score by the number of questions completed; increase in total score is associated with decreased quality of life and increased symptom burden
12-Item Short Form Survey (SF-12) | 5 Minutes
  The SF-12 is a self-reported outcome measure .The questionnaire developed to evaluate health-related quality of life, physical function (2 items), physical role limitation (2 items), pain (1 item), general health (1 item), energy (1 item), social function (1 item) It consists of 8 sub-dimensions and 12 items, including emotional role restriction (2 items) and mental health (2 items). The score that can be obtained from the scale varies between 0 and 100, and a higher score is an indicator of better health-related quality of life.
PHYSICAL ACTIVITY SCALE-2 | 5 Minutes
  It is used to determine the daily and weekly physical activity levels of adults. The scale consists of 9 items that measure sedentary behavior at work, transportation and leisure time and physical activity levels of different intensities (light, moderate and vigorous). The daily and weekly physical activity level of the person can be estimated by using the metabolic equivalent (MET) equivalent of each item asked in the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Raziye Şavkın, Assoc. Prof., Study Chair — Pamukkale University; Ömer Faruk Can, PT, Principal Investigator — Pamukkale University; Ufuk Kutluana, Assoc. Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No